CLINICAL TRIAL: NCT03063216
Title: Visual Outcome Evaluation and Genetic Analysis: Shanghai Pediatric Cataract Study
Brief Title: Shanghai Pediatric Cataract Study
Status: Recruiting | Type: Observational
Sponsor: Evidence Based Cataract Study Group (Other)
Collaborators: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: SH-PCS
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Cataract; Congenital Cataract; Traumatic Cataract; Visual Outcome; Genetic Anticipation
MeSH Terms: conditions — Anticipation, Genetic | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Samples of blood, aqueous humor, anterior capsular membranes and lens tissues from pediatric cataract patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Congenital cataract group: Cataract patients diagnosed with congenital cataract.
  Interventions: Procedure: intraocular lens implantation
- Traumatic cataract group: Cataract patients diagnosed with traumatic cataract.
  Interventions: Procedure: intraocular lens implantation

INTERVENTIONS:
Procedure: intraocular lens implantation — 1）Pediatric cataract patients with intraocular lens implantation and those without intraocular lens implantation；2）Traumatic cataract patients with intraocular lens implantation and those without intraocular lens implantation

SUMMARY:
The purpose of this study is to evaluate the long-term visual outcome of the cataract surgery using a large-scale and comprehensive database of pediatric cataract participants, including congenital and traumatic cataract. The investigators will further investigate into the various genetic and environmental factors that may contribute to the pathogenesis of pediatric cataract.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pediatric cataract
* Must be able to cooperate with the ophthalmic examination

Exclusion Criteria:

* Clinical diagnosis of mental illness
* Mentally disabled

Ages: 2 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Medical centre: Eye and ENT Hospital of Fudan University
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2045-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the visual outcomes of pediatric cataract patients. | Follow-up until ten years after surgery.
  Visual outcomes are evaluated including visual acuity with or without correction, refractive changes, intraocular pressure, fundus function, fixation type, vision development, growth of axial length, contrast sensitivity and other visual outcome measurements.
Genetic diversity based on biospecimen samples of pediatric cataract patients. | Analyzed within six months after surgery.
  Sequencing of genes (including exons, promoters, 5' UTR and 3' UTR sequences) on a large scale to intensively investigate into the sites and functions of single nucleotide polymorphism (SNP) correlated with clinical features of congenital cataract patients, compared to traumatic cataract patients.Samples of blood, aqueous humor, anterior capsular membranes and lens tissues were applied for the genetic analysis.

SECONDARY OUTCOMES:
Differences in the clinical phenotypes of pediatric cataract patients. | Evaluated before receiving the cataract surgery.
  Cataract type and severity of ametropic cataract patients are evaluated and images are captured before receiving the cataract surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, M.D., Study Chair — Eye and ENT Hospital of Fudan University; Xiangjia Zhu, M.D., Study Director — Eye and ENT Hospital of Fudan University; Keke Zhang, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University; Wenwen He, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University; Yu Du, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University; Yinglei Zhang, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University; Ruiqi Chang, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu X, He W, Du Y, Kraus CL, Xu Q, Sun T, Yu J, Lu Y. Presence of Posterior Staphyloma in Congenital Cataract Children. Curr Eye Res. 2019 Dec;44(12):1319-1324. doi: 10.1080/02713683.2019.1637437. Epub 2019 Jul 5. PMID 31246115